CLINICAL TRIAL: NCT01196208
Title: An Open-label, Treatment-option Protocol of Brentuximab Vedotin in Patients With Relapsed or Refractory Hodgkin Lymphoma, Systemic Anaplastic Large Cell Lymphoma, or CD30-positive Cutaneous T-cell Lymphoma
Brief Title: A Treatment-Option Protocol to Provide Brentuximab Vedotin to Eligible Patients Completing Studies SGN35-005 or C25001
Status: No longer available | Type: Expanded Access
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SGN35-010; 2010-020363-21 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous
Keywords: Disease, Hodgkin; Lymphoma; Monomethylauristatin E; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Non-Hodgkin; Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Hematologic Diseases; Immunotherapy
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Lymphoma; Hematologic Diseases | interventions — Brentuximab Vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — Every 21 days by intravenous infusion (1.8 mg/kg)
  Other Names: SGN-35

SUMMARY:
The purpose of this study is to provide the option of brentuximab vedotin treatment to eligible patients in studies SGN35-005 and C25001

DETAILED DESCRIPTION:
The protocol was amended to reflect the change from a phase 2/3 to a study with an expanded access program (EAP) in the US that would include patients with ALCL and HL. A later amendment allowed patients with CD30-positive cutaneous T-cell lymphoma to enroll. Enrollment may continue and patients may receive brentuximab vedotin treatment on study until the drug is commercially approved and available to patients in a geographic region.

ELIGIBILITY:
Inclusion Criteria:

* Participated in either the SGN35-005 or C25001 clinical study and experienced progression. Patients who received brentuximab vedotin in C25001 must have had an objective response at the time of discontinuation.
* Completed any previous treatment with radiation, chemotherapy, biologics and/or investigational agents at least 4 weeks prior to the first dose of brentuximab vedotin

Exclusion Criteria:

* History of another primary malignancy that has not been in remission for at least 3 years
* Known cerebral/meningeal disease
* Peripheral neuropathy of grade 2 or greater
* Females who are pregnant or breastfeeding

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Liga Ulmane, MD, Study Director — PSI Company Ltd.
Locations (31):
- United States (3):
  - Stanford Cancer Center, Stanford, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
- Peter MacCallum Cancer Center, Melbourne, Australia
- Leuven University Hospital, Leuven, Belgium
- Bulgaria (2):
  - Specializirana bolnica aktivno lechenie detsa ohcohematologichni zabolyavania Hematologichno, Sofia
  - Specializirana bolnica za aktivno lechenie na hematologichni zabolyavania, Sofia
- France (3):
  - Hopital Saint-Louis/Service d'Hematologie, Paris, Cedex 10
  - South Lyon Hospital Center, Department of Dermatology, Lyon
  - Centre Henri Becquerel / Centre Regional de Lutte Contre le Cancer, Rouen
- Johannes Wesling Hospital Minden, Department of Dermatology, Minden, Germany
- Hungary (3):
  - Szent Istvan es Szent Laszlo Korhaz Rendelointezet Haematologiai es Ossejt-transzplantacios osztaly, Budapest
  - Debreceni Egyetem Orvos és Egeszsegtudomanyi Centrum, III. sz. Belgyogyaszati Klinika, Debrecen
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikat Kozpont, Szeged
- Italy (2):
  - Polyclinic S. Orsola-Malpighi, Institute of Hematology and Medical Oncology "Lorenzo and Ariosto Seragnoli", Bologna
  - IRCCS University Hospital San Martino, Genoa
- Poland (3):
  - Klinika Hematologii, Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Klinika Hematologii, Instytut Hematologii i Transfuzjologii, Warsaw
  - Centrum Onkologii Institut im. Marii Sklodowskiej-Curie, Warsaw
- Romania (3):
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Sectia Clinica Hematologie si Transplant Medular, Târgu Mureş, Mureș County
  - Fundeni Clinical Institute, Center for Hematology and Bone Marrow Transplantation, Bucharest
  - Institutul Clinic Fundeni, Centrul de Hematologie si Transplant Medular Stefan Berceanu, Bucharest
- Russia (4):
  - Rossijskij onkologicheskij nauchnyj centr im. N.N. Blokhina RAMN, Moscow
  - Gematologicheskj nauchnyj centr RAMN, Moscow
  - Research Institute of Clinical Immunology, Novosibirsk
  - Sankt-Peterburgskij gosudarstvennyj medicinskij universitet im. akademika I. P. Pavlova, Saint Petersburg
- Clinical Center of Serbia, Clinic of Hematology, Belgrade, Serbia
- University Hospital 12 de Octubre, Department of Dermatology, Madrid, Spain
- University Hospital Zurich, Department of Dermatology, Zurich, Switzerland
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - St John's Institute of Dermatology, London